CLINICAL TRIAL: NCT04178473
Title: Total Versus Subtotal Abdominal Hysterectomy at Time of Abdominal Sacrocolpopexy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Mohammad Abdel-Rahman Mohammad Ahmed, Doctor, South Valley University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: OBGYN 0101
Record Dates: First submitted 2019-11-24; First posted 2019-11-26 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Prolapse Genital
Keywords: hysterectomy; sacrocolpopexy

STUDY DESIGN:
Intervention Model Description: Group A will have total abdominal hysterectomy Group B will have subtotal abdominal hysterectomy Sacrocolpopexy will be done using Polypropylene mesh for all women with uterovaginal prolapse
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double (Participant, Investigator) closed envelop will be used for randomization. The patient and the investigator will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- total abdominal hysterectomy (Active Comparator): Total abdominal hysterectomy at the time of sacrocolpopexy operation for uterovaginal prolapse
  Interventions: Procedure: total abdominal hysterectomy
- subtotal abdominal hysterectomy (Active Comparator): subtotal abdominal hysterectomy at the time of sacrocolpopexy operation for uterovaginal prolapse
  Interventions: Procedure: Subtotal abdominal hysterectomy

INTERVENTIONS:
Procedure: total abdominal hysterectomy — total abdominal hysterectomy at time of sacrocolpopexy
  Arms: total abdominal hysterectomy
Procedure: Subtotal abdominal hysterectomy — Subtotal abdominal hysterectomy at time of sacrocolpopexy
  Arms: subtotal abdominal hysterectomy

SUMMARY:
Uterovaginal prolapse is a common disease. Due to high failure rate that occur following vaginal hysterectomy, sacrocolpopexy is investigated by many resarchers to manage uterovaginal prolapse in non-hystrectomized women.

In this study the investigator will compare the result of total versus subtotal hysterectomy at the time of sacrocolpopexy.

Study design: Randomized controlled trial

Intervention:

Group A will have total abdominal hysterectomy Group B will have subtotal abdominal hysterectomy

DETAILED DESCRIPTION:
Uterovaginal prolapse is a common disease. Sacrocolpopexy is essentially invented to manage prolapse of the vault following hysterectomy. Due to high failure rate that occur following vaginal hysterectomy, sacrocolpopexy is investigated by many resarchers to manage uterovaginal prolapse in non-hystrectomized women. The main drawback of sacrocolpopexy is the risk of mesh erosion. The incidence of mesh erosion is 0-5% at follow up of 1 year and 0.5% at follow up of 7 years. After total hysterectomy, the mesh is sutured to the vaginal wall using non-absorbable sutures. Sutures that span the whole thickness of vaginal and involve the vaginal skin was considered the probable factor that result in mesh erosion. After subtotal hysterectomy, the mesh is fixed to the anterior and the posterior cervical surfaces. The cervix has thick wall and the risk associated with "deep" stiches does not exist.

In this study the investigator will compare the result of total versus subtotal hysterectomy at the time of sacrocolpopexy.

Patients and methods

Study design:

Randomized controlled trial

Patients:

Data will be collected from the patients admitted to the obstetrics and gynecology department, Qen faculty of medicine, South Valley University, Egypt from the 1st of January 2019 until 30th of December 2019. Follow up data will be collected until 30th of December 2020. Written consent will be obtained at time of recruitment. The Inclusion criteria are nonhystrectomized patients who will undergo sacrocolpopexy. Exclusion criteria were (1) women age less than 40; (2) desire to retain the uterus; (3) women who are unfit for lengthy surgery. Randomization will be through closed envelop method.

Intervention Group A will have total abdominal hysterectomy Group B will have subtotal abdominal hysterectomy Sacrocolpopexy will be done using Polypropylene mesh. Both groups will be done by the same surgeon using the following technique: dissection of the vesicovaginal and the rectovaginal spaces to prepare for the site of mesh placement. Dissection will be continued in the rectovaginal septum using sharp and blunt dissection until reaching the level of the levator ani (the length of the posterior vaginal mesh arm is nearly equal to the total vaginal length). The limit of the dissection in the vesicovaginal plane is down to the bladder neck (known by palpation of the Foley's catheter balloon) after lateralization of the ureters. The mesh is sutured to the anterior and the posterior vaginal wall the mesh using non-absorbable sutures. In women with subtotal hysterectomy, the mesh will be also sutured to the cervix. The mesh is then sutured to the anterior longitudinal ligament on the anterior surface of the fifth lumbar vertebra and the sacral promontory using non-absorbable sutures. Suturing of the peritoneum over the mesh will be done.

Outcomes:

The primary outcome will be mesh erosion. Secondary outcomes will be complications including recurrence

ELIGIBILITY:
Inclusion Criteria:

* nonhystrectomized patients who will undergo sacrocolpopexy for uterovaginal prolapse

Exclusion Criteria:

* women age less than 40
* desire to retain the uterus
* women who are unfit for lengthy surgery

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — nonhystrectomized patients who will undergo sacrocolpopexy for uterovaginal prolapse
Enrollment: 70 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
Mesh erosion | 12 months or more
  Mesh exposure through the lumen of the vagina, bladder, or rectum

SECONDARY OUTCOMES:
recurrence | 12 months or more
  recurrence of vaginal wall prolapse or vault prolapse

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad AM Ahmed, MD, Principal Investigator — South Valley University, Qena Faculty of Medicine, Obstetrics and Gynecology Department, Qena, Qena, Egypt
Locations (1):
- South Valley University, Qena Faculty of Medicine, Obstetrics and Gynecology Department, Qina, Qena Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared in unanonomous manner with the predetermined group of researchers
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: throughout the period of research until end of the study
Access Criteria: IPD will be shared with the predetermined group of researchers as accepted by the local ethical and research committee.

REFERENCES:
- [Background] Barrington JW, Edwards G. Posthysterectomy vault prolapse. Int Urogynecol J Pelvic Floor Dysfunct. 2000;11(4):241-5. doi: 10.1007/s001920070033. PMID 11005477
- [Background] Cayrac M, Warembourg S, Le Normand L, Fatton B. [Does hysterectomy modifies the anatomical and functional outcomes of prolapse surgery?: Clinical Practice Guidelines]. Prog Urol. 2016 Jul;26 Suppl 1:S73-88. doi: 10.1016/S1166-7087(16)30430-4. French. PMID 27595628
- [Background] Coolen AWM, Bui BN, Dietz V, Wang R, van Montfoort APA, Mol BWJ, Roovers JWR, Bongers MY. The treatment of post-hysterectomy vaginal vault prolapse: a systematic review and meta-analysis. Int Urogynecol J. 2017 Dec;28(12):1767-1783. doi: 10.1007/s00192-017-3493-2. Epub 2017 Oct 16. PMID 29038834
- [Background] Cundiff GW, Varner E, Visco AG, Zyczynski HM, Nager CW, Norton PA, Schaffer J, Brown MB, Brubaker L; Pelvic Floor Disorders Network. Risk factors for mesh/suture erosion following sacral colpopexy. Am J Obstet Gynecol. 2008 Dec;199(6):688.e1-5. doi: 10.1016/j.ajog.2008.07.029. Epub 2008 Oct 31. PMID 18976976
- [Background] Ismail S, Duckett J, Rizk D, Sorinola O, Kammerer-Doak D, Contreras-Ortiz O, Al-Mandeel H, Svabik K, Parekh M, Phillips C. Recurrent pelvic organ prolapse: International Urogynecological Association Research and Development Committee opinion. Int Urogynecol J. 2016 Nov;27(11):1619-1632. doi: 10.1007/s00192-016-3076-7. Epub 2016 Jul 5. PMID 27379891